CLINICAL TRIAL: NCT02164578
Title: Microvascular and Antiinflammatory Effects of Rivaroxaban Compared to Low Dose Aspirin in Type-2 Diabetic Patients With Very High Cardiovascular Risk and Subclinical Inflammation
Brief Title: Microvascular and Antiinflammatory Effects of Rivaroxaban Compared to Aspirin in Type-2 Diabetic Patients With Subclinical Inflammation and High Cardiovascular Risk
Acronym: MicroVasc-DIVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MicroVasc-DIVA
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetic Patients
MeSH Terms: interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivaroxaban (Experimental): 5mg b.i.d. for 20 weeks (primary phase) + additional 32 weeks (extension phase)
  Interventions: Drug: Rivaroxaban
- Aspirin (Active Comparator): 100mg once daily for 20 weeks (primary phase) + additional 32 weeks (extension phase)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Rivaroxaban
  Arms: Rivaroxaban
Drug: Aspirin
  Arms: Aspirin

SUMMARY:
Study to investigate microvascular and antiinflammatory effects of Rivaroxaban compared to low dose aspirin in type 2 diabetic patients.

Especially patients with cardiovascular disease and subclinical inflammation are in the focus of interest.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes duration between 2 and 20 years
* Two or more components of metabolic syndrome:

  * HDL-cholesterol < 1.0 mmol/L (in males) or < 1.3 mmol/L (in females)
  * Elevated triglycerides (> 1.7 mmol/L)
  * Elevated blood pressure (> 130 mmHg systolic and/or >85 mmHg diastolic or antihypertensive treatment)
  * Elevated waist circumference (> 102 cm in males, > 85 cm in females)
* Or at least one of the following

  * Carotid ultrasound showing an IMT > 1 mm and plaque of carotid artery or
  * Left ventricular hypertrophy or
  * Increased UACR in the absence of other renal diseases than diabetic nephropathy
* Increased hsCRP (> 2 mg/l but < 10 mg/l) at or within 6 months prior to screening and/or increased PAI 1 (> 15 ng/ml) at or within 6 months prior to screening (the historical hsCRP or PAI 1 value can be used only if the patient was in stable conditions regarding the concomitant diseases and statin therapy since the time point of measurement)
* Stable treatment with statins (if tolerated/clinically indicated)
* Age 40 - 75 years

Exclusion Criteria:

* Major cardiovascular (CV) event with need for oral anticoagulation or platelet inhibitor therapy or acute coronary syndrome < 12 month before study entry
* Sustained uncontrolled hypertension: systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg
* Hypersensitivity to the active substance or to any of the excipients
* Active clinically significant bleeding
* Lesion or condition, if considered to be a significant risk for major bleeding
* Concomitant treatment of acute coronary syndrome (ACS) with antiplatelet therapy in patients with a prior stroke or a transient ischemic attack (TIA)
* Hepatic disease associated with coagulopathy and clinically relevant bleeding risk including cirrhotic patients with Child Pugh B and C
* Chronic renal failure with eGFR < 15 ml/min (MDRD formula)
* Pregnant or breast-feeding woman and woman without adequate method of contraception.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pistrosch, Dr. med., Principal Investigator — GWT-TUD GmbH
Locations (5):
- Germany (5):
  - Krankenhaus Dresden-Friedrichstadt, Dresden, Saxony
  - Universitätsmedizin Berlin / Charité Campus Buch, Berlin
  - Gemeinschaftspraxis Dr. Schaper/ Dr. Faulmann, Dresden
  - GWT-TUD GmbH / Studienzentrum Hanefeld, Dresden
  - Cardiologicum Prina, Pirna

REFERENCES:
- [Derived] Pistrosch F, Matschke JB, Schipp D, Schipp B, Henkel E, Weigmann I, Sradnick J, Bornstein SR, Birkenfeld AL, Hanefeld M. Rivaroxaban compared with low-dose aspirin in individuals with type 2 diabetes and high cardiovascular risk: a randomised trial to assess effects on endothelial function, platelet activation and vascular biomarkers. Diabetologia. 2021 Dec;64(12):2701-2712. doi: 10.1007/s00125-021-05562-9. Epub 2021 Sep 8. PMID 34495376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 14th Apr 2015 through 21st Dec 2017, a total of 239 patients were screened at 4 study sites in Germany. Of them, 60 patients did not meet the eligibility criteria. 188 patients were planned to enrol and 80 patients of them should included in the extension period of the study.
Pre-assignment Details: 179 patients were randomized to one of the two treatment groups, 89 to receive rivaroxaban and 90 to receive acetylsalicylic acid (ASA). In total, 73 patients were included in the extension period, 37 of them received rivaroxaban and 36 received ASA.
Groups:
- Rivaroxaban: 5mg b.i.d. for 20 weeks (treatment phase) + additional 32 weeks (extension phase)
- Aspirin: 100mg once daily for 20 weeks (treatment phase) + additional 32 weeks (extension phase)
Period: Treatment Period
Arm/Group | Rivaroxaban | Aspirin
Started | 89 | 90
Completed | 72 | 79
Not Completed | 17 | 11
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 13 | 6
Not completed — Early termination due to expiry of study medication | 1 | 0
Not completed — Protocol Violation | 0 | 2
Period: Extension Period
Arm/Group | Rivaroxaban | Aspirin
Started (According to protocol only 80 patients were planned to participate in the extion period. In total, 73 subjects were included in the extension period.) | 37 (37 of 40 planned patients continued treatment period and were included in the extension period) | 36 (36 of 40 planned patients continued treatment period and were included in the extension period)
Completed | 30 | 35
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Expiry of study medication | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed for the full analysis set (n=179)
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Aspirin | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Continuous [Mean (Full Range); unit: years] | 64.2 [40 to 76] | 64.7 [45 to 76] | 64.4 [40 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 44 | 95
  Male | 38 | 46 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 89 | 90 | 179
Region of Enrollment [Number; unit: participants]
  Germany | 89 | 90 | 179
BMI [Mean (Full Range); unit: kg/m^2] | 33.2 [24 to 55] | 33.4 [25 to 47] | 33.3 [24 to 55]
Duration of diabetes [Mean (Full Range); unit: years] | 9.21 [2 to 28] | 9.24 [2 to 20] | 9.22 [2 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-ischemic Forearm Blood Flow
Description: Change of maximal postischemic forearm blood flow during reactive hyperaemia after 5 min of forearm ischemia (FBF max. ml/100ml).
  Difference of change in post-ischemic forearm blood flow measured by venous occlusion plethysmography at baseline and after 20 weeks treatment with rivaroxaban or aspirin.
Time Frame: Baseline and week 20
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ml/100ml
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 83 | 84
ml/100ml | 3.60 (4.69) | 1.00 (5.27)
Statistical Analysis 1: Comparison: Rivaroxaban vs Aspirin; The hypothesis H0 is tested against the one-sided alternative hypothesis H1 H0: µ∆FBF,Riva, week 20 ≤ µ∆FBF, ASA, week 20 versus H1: µΔFBF, Riva, week 20 > µΔFBF, ASA, week 20 by test procedures for continuous data; Test type: Superiority; p = 0.004, ANCOVA; ANCOVA for repeated measurements with baseline as covariate

2. Primary Outcome: Change in Pulse Wave Velocity
Description: Change in pulse wave velocity as a marker of arterial stiffness (measured by IEM Mobil-O-Graph)
Time Frame: Baseline and week 52
Population: Full Analysis Set of the extension phase
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 34 | 36
m/s | 0.24 (0.62) | 0.51 (0.57)
Statistical Analysis 1: Comparison: Rivaroxaban vs Aspirin; Test type: Other; p = 0.070, ANCOVA

3. Secondary Outcome: Change in Post-ischemic Forearm Blood Flow
Description: Difference of change in post-ischemic forearm blood flow measured by venous occlusion plethysmography at baseline and after 52 weeks treatment with rivaroxaban or aspirin.
Time Frame: Baseline and week 52
Population: Full Analysis Set of the extension phase
Measure: Mean (Standard Deviation); unit: ml/100ml
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 29 | 30
ml/100ml | 6.11 (8.83) | 1.56 (5.34)
Statistical Analysis 1: Comparison: Rivaroxaban vs Aspirin; Test type: Other; p = 0.045, ANCOVA; ANCOVA for repeated measurements with baseline as covariate

4. Secondary Outcome: Change in Pulse Wave Velocity
Description: Change in pulse wave velocity as a marker for arterial stiffness (measured by IEM Mobil-O-Graph)
Time Frame: Baseline to week 20
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 82 | 85
m/s | 0.02 (0.44) | 0.14 (0.53)
Statistical Analysis 1: Comparison: Rivaroxaban vs Aspirin; Test type: Other; p = 0.125, ANCOVA

5. Secondary Outcome: Change in Skin Blood Flow
Description: Change in skin blood flow for assessment of peripheral skin microcirculatory function (measured by laserdopplerfluxmetry; LDF)
Time Frame: Baseline to week 20
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 76 | 79
arbitrary units | 3.47 (44.7) | -6.01 (34.0)
Statistical Analysis 1: Comparison: Rivaroxaban vs Aspirin; Test type: Other; p = 0.217, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Skin Blood Flow
Description: as for outcome 5
Time Frame: Baseline to week 52
Population: Full Analysis Set of the extension phase
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 34 | 36
arbitrary units | -7.3 (45.1) | 5.8 (59.5)
Statistical Analysis 1: Comparison: Rivaroxaban vs Aspirin; Test type: Other; p = 0.589, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Major Bleeding
Description: Major bleeding defined as clinically overt and associated with one of the following: 1) reduction of hemoglobin level of 2 g/L or 2) required transfusion of at least 2 units of red cells or, involved a critical organ or was fatal, in accordance with the recommendation of the International Society on Thrombosis and Hemostasis (ISTH).
Time Frame: Week 1 to week 20
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 89 | 90
events | 1 | 0

8. Secondary Outcome: Major Bleeding
Description: as for outcome 7
Time Frame: Week 1 to week 52
Population: Safety Analysis Set of the extension phase
Measure: Number; unit: events
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 37 | 36
events | 0 | 0

9. Secondary Outcome: Clinically Relevant Non-major (CRNM) Bleeding
Description: Clinically relevant non-major (CRNM) bleeding defined as at least one of the following:
  * spontaneous skin hematoma of at least 25 cm
  * spontaneous nose bleeding of more than 5 minutes duration
  * macroscopic hematuria, either spontaneous or, if associated with an intervention, lasting more than 24 hours
  * spontaneous rectal bleeding (more than spotting on toilet paper)
  * gingival bleeding for more than 5 minutes
  * bleeding leading to hospitalization and/or requiring surgical treatment
  * bleeding leading to a transfusion of less than 2 units of whole blood or red cells
  * any other bleeding event considered clinically relevant by the investigator
Time Frame: Week 1 to week 20
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 89 | 90
events | 11 | 1

10. Secondary Outcome: Clinically Relevant Non-major (CRNM) Bleeding
Description: as for outcome 9
Time Frame: Week 1 to week 52
Population: Safety Analysis Set of the extension phase
Measure: Number; unit: events
Arm/Group | Rivaroxaban | Aspirin
Number analyzed (Participants) | 37 | 36
events | 6 | 1

ADVERSE EVENTS:
Time Frame: Randomization to Week 20 (primary phase) and to Week 52 (extension phase)
Arm/Group | Rivaroxaban | Aspirin
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 4/89 | 6/90
Other Adverse Events (participants affected / at risk) | 0/89 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (N=89) | Aspirin (N=90)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02164578/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02164578/SAP_001.pdf